CLINICAL TRIAL: NCT02935062
Title: New Therapeutical Perspectives in Cases of Phonological Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Santa Maria (Other)
Responsible Party: Principal Investigator, Marcia Keske Soares, Professora Doutora, Universidade Federal de Santa Maria
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 28053914.1.0000.5346
Record Dates: First submitted 2016-09-15; First posted 2016-10-17 (Estimated); Results first posted 2019-12-18 (Actual); Last update posted 2019-12-18 (Actual); Status verified 2019-11

CONDITIONS: Speech Sound Disorders
Keywords: Speech; Speech Therapy; Speech Sound Disorders; Phonological Disorders; Auditory Perception
MeSH Terms: conditions — Speech Sound Disorder; Speech; Communication Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Traditional Phonological Therapy (Active Comparator): This intervention will be intermediated by the traditional model cycles. This approach has the principle of treating the suppression of operant phonological processes in child's speech, from the awareness of sound-target characteristics operating in that phonological process.
  Interventions: Behavioral: Traditional Phonological Therapy
- Software Phonological Therapy- SIFALA (Experimental): This intervention will be intermediated by the software SIFALA. The software SIFALA, allows to select target segments using the Modelo de Estratos (second model Strata), based on the level segment of production and complexity of distinctive features, from the child's sound system analysis and planned generalizations. It also seeks the treatment of phonological disorders, by selection stimulus words in more favorable environments and playful activities with computer resource for the correct production of the target segment in the words stimulus, promoting the spread segments.
  Interventions: Behavioral: Software Phonological Therapy- SIFALA
- Placebo Therapy (Placebo Comparator): No interventional group. This group will be the sham group. The proposed activities will be fun games on the computer, there is no relationship with speech and it will be not emphasized the correct sound production, will only play activities.
  Interventions: Behavioral: Placebo Therapy

INTERVENTIONS:
Behavioral: Traditional Phonological Therapy — Phonological therapy based on generalizing the sounds presented by figures, repetition and naming words.
  Arms: Traditional Phonological Therapy
Behavioral: Software Phonological Therapy- SIFALA — The phonological thearapy of this group will be based on software use with phonological model already developed, using naming and repetition of sounds.
  Arms: Software Phonological Therapy- SIFALA
Behavioral: Placebo Therapy — No intervention to improve speech.
  Arms: Placebo Therapy

SUMMARY:
The aim of this study is to verify phonological and auditory aspects of children submitted to traditional phonological therapy, phonological therapy using a software and placebo therapy in children with phonological disorders.

DETAILED DESCRIPTION:
The study will provide different therapeutic approaches for cases of phonological disorders, the classical approach would be mediated by Cycles Model, innovated approach is performed by means of an intervention speech software-SIFALA, there will still be the group that does not receive any of the proposals therapies that will be the placebo group.The study will provide 25 sessions for each group, with 30 minutes in each group. At the end of these sessions, the placebo group will receive one of the therapeutic approaches. With these three study groups, the investigators understand in what manner to obtain correct sounds is more effective.

ELIGIBILITY:
Inclusion Criteria:

* Parents/guardians and child agree to participate and have signed the Informed Consent Form;
* Have age between 4:0 to 8:11 (years:months);
* Present diagnosis of phonological disorders;
* Present hearing thresholds within the normal range

Exclusion Criteria:

* Present neurological impairment, emotional and/or cognitive clearly diagnosed, or have complaint;
* Present any degree of hearing loss is the type conductive, mixed or sensorineural, and middle ear disorders in time of selection, as well as having presented otitis complaints;
* Present language impairment associated with speech sound disorder;
* Present commitment in the stomatognathic system that can interfere in the speech production;
* Have been received speech and language therapy before.

Ages: 4 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2016-07; Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marcia Keske-Soares, PhD, Study Director — Universidade Federal de Santa Maria
Locations (2):
- Brazil (2):
  - Universidade Federal de Santa Maria- campus Camobi e centro- Floriano Peixoto 1709., Santa Maria, Rio Grande do Sul
  - Federal University of Santa Maria, Santa Maria, Rio Grande do Sul

IPD SHARING:
Plan to Share IPD: Yes
The plan to make the individual data available is in accordance with the criteria adopted in the research and the research ethics committee of the educational institution, which developed the study.
  The results, placed on the platform of this randomized clinical trial, can be used by other researchers.
Supporting Information: ICF
Time Frame: Results were exposed for three years
Access Criteria: Researchers with access to Clinical Trials and those who wish to contact the responsible researcher.

RESULTS

PARTICIPANT FLOW:
Groups:
- Traditional Phonological Therapy- CYCLES: This intervention will be intermediated by the traditional model cycles. This approach has the principle of treating the suppression of operant phonological processes in child's speech, from the awareness of sound-target characteristics operating in that phonological process.
  Traditional Phonological Therapy: Phonological therapy based on generalizing the sounds presented by figures, repetition and naming words.
Period: Overall Study
Arm/Group | Software Phonological Therapy- SIFALA | Traditional Phonological Therapy- CYCLES | Placebo Therapy
Started | 8 | 8 | 8
Completed | 8 | 8 | 8
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Software Phonological Therapy- SIFALA | Traditional Phonological Therapy- CYCLES | Placebo Therapy | Total
Number analyzed (Participants) | 8 | 8 | 8 | 24
Age, Continuous [Mean (Full Range); unit: years] | 7.81 [5.1 to 8.1] | 7.48 [6.2 to 7.5] | 6.51 [4.9 to 8.1] | 7.26 [4.0 to 8.1]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 2 | 10
  Male | 4 | 4 | 6 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 2 | 3
  White | 7 | 8 | 6 | 21
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Brazil | 8 | 8 | 8 | 24

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Consonants Correct (PCC) Pre-treatment and Post-treatment Phonological Instrument
Description: The percentage of correct consonants corresponds to the number of phonemes produced by the child, evaluated initially before starting treatment and at the end of treatment. The variable of this calculation is based on the percentage which is determined at what phonological level of disorder the child is at. It is expected that at the end of treatment the percentage of correct consonants will increase due to the therapy stimuli offered.
Time Frame: 10 weeks
Population: The population is described by the age and using the variables of PCC, phonemes acquired The numbers shows the meand and standard deviation after the treatment.
Measure: Mean (Standard Deviation); unit: PCC - (%)
Groups:
- Ciclos- Therapy: This intervention will be intermediated by the traditional model cycles. This approach has the principle of treating the suppression of operant phonological processes in child's speech, from the awareness of sound-target characteristics operating in that phonological process.
  Traditional Phonological Therapy: Phonological therapy based on generalizing the sounds presented by figures, repetition and naming words.
Arm/Group | Ciclos- Therapy | Software Phonological Therapy- SIFALA | Placebo Therapy
Number analyzed (Participants) | 8 | 8 | 8
PCC - (%)
  PCC Pre-treatment | 70.63 (17.77) | 68.13 (12.53) | 75.5 (8.60)
  PCC Pos-treatment | 79.88 (19.86) | 80.63 (14.11) | 82.88 (10.68)
Statistical Analysis 1: Comparison: Ciclos- Therapy vs Software Phonological Therapy- SIFALA vs Placebo Therapy; Test type: Superiority; p = 0.001, t-test, 1 sided

2. Primary Outcome: P300- Long-latency Auditory Evoked Potential
Description: Electrophysiological evaluation of the auditory pathway through the protocol, Pretreatment and Post-treatment P300 waves were analyzed by the latency according to the parameters of MacPherson (1996).
  The electrophysiological protocol was performed before and after therapy. The marking of the waves was judged by specialist judges in the field of audiology.
  The variable that predicts P300 latency is quantified in milliseconds (ms
Time Frame: 10 weeks.
Population: The same sample was evaluated with this P300 variable, quantified in milliseconds (ms), which corresponds to the P300 electrophysiological wave latency.
Measure: Mean (Standard Deviation); unit: (ms) milliseconds
Arm/Group | Ciclos- Therapy | Software Phonological Therapy- SIFALA | Placebo Therapy
Number analyzed (Participants) | 8 | 8 | 8
(ms) milliseconds
  P300- Pre-Treatment | 383.60 (25.15) | 373.28 (50.45) | 357.33 (10.21)
  P300- Pos-Treatment | 344.00 (20.09) | 362.66 (29.67) | 353.23 (29.15)
Statistical Analysis 1: Comparison: Ciclos- Therapy vs Software Phonological Therapy- SIFALA vs Placebo Therapy; Test type: Superiority; p = 0.011, t-test, 1 sided

ADVERSE EVENTS:
Time Frame: 10 weeks
Description: No adverse events, fortunately, were observed during the research.
Arm/Group | Software Phonological Therapy- SIFALA | Traditional Phonological Therapy- CYCLES | Placebo Therapy
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8

LIMITATIONS AND CAVEATS:
Limitations:

Small number of the sample, since the study requires treatment, so there are few researchers for the treatments. Also some limitations regarding the human subjectivity of results. However the participants adhered to the treatment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-20): https://cdn.clinicaltrials.gov/large-docs/62/NCT02935062/Prot_SAP_000.pdf